CLINICAL TRIAL: NCT01335724
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Parallel Group Phase IV Study to Evaluate the Efficacy and Safety of Diclofenac 1.16% Gel in Subjects With Acute Neck Pain
Brief Title: Efficacy and Safety of Diclofenac 1.16% Gel in Subjects With Acute Neck Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 862-P-201
Record Dates: First submitted 2011-04-13; First posted 2011-04-14 (Estimated); Results first posted 2012-07-18 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-06

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — diclofenac diethylamine; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diclofenac diethylamine 1.16% gel (Experimental)
  Interventions: Drug: Diclofenac diethylamine 1.16% gel
- placebo gel (Placebo Comparator)
  Interventions: Drug: Placebo gel

INTERVENTIONS:
Drug: Diclofenac diethylamine 1.16% gel — Diclofenac diethylamine 1.16% gel
  Arms: Diclofenac diethylamine 1.16% gel
Drug: Placebo gel — Placebo gel
  Arms: placebo gel

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of diclofenac 1.16% gel compared with placebo applied four times a day in subjects with acute neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, age range 18 and over.
* Patient with acute neck pain meeting baseline pain intensity level and duration

Exclusion Criteria:

* Pain medication was taken within the 6 hours that precede randomization.
* Patient with chronic neck pain as defined as pain for 3 months or longer
* Any neck pain that is attributable to any organic disease, such as prolapsed disc, spondylolisthesis, osteomalacia, inflammatory arthritis, metabolic, neurological diseases or tumors.
* Any recent strains of the neck muscles documented by the clinical evaluation and anamnesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - NCH investigative site, Cologne
  - NCH investigative site, Essen
  - NCH investigative site, Munich

REFERENCES:
- [Derived] Predel HG, Giannetti B, Pabst H, Schaefer A, Hug AM, Burnett I. Efficacy and safety of diclofenac diethylamine 1.16% gel in acute neck pain: a randomized, double-blind, placebo-controlled study. BMC Musculoskelet Disord. 2013 Aug 21;14:250. doi: 10.1186/1471-2474-14-250. PMID 23964752

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diclofenac Diethylamine 1.16% Gel | Placebo Gel
Started | 36 | 36
Completed | 36 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diclofenac Diethylamine 1.16% Gel | Placebo Gel | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 34 | 70
  >=65 years | 0 | 2 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 29.8 (10.5) | 37.8 (15.2) | 33.8 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 14 | 33
  Male | 17 | 22 | 39
Region of Enrollment [Number; unit: participants]
  Germany | 36 | 36 | 72

OUTCOME MEASURES:

1. Primary Outcome: Pain on Movement
Description: Pain on movement on a 100 mm visual analog scale. Minimum score =0 mm "no pain". Maximum score =100 mm "extreme pain".
Time Frame: 48 h
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac Diethylamine 1.16% Gel | Placebo Gel
Number analyzed (Participants) | 36 | 36
mm | 19.5 (12.9) | 56.9 (16.1)

2. Secondary Outcome: Pain at Rest
Description: Pain at Rest on a 100 mm visual analog scale. Minimum score =0 mm "no pain". Maximum score =100 mm "extreme pain".
Time Frame: 96h
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac Diethylamine 1.16% Gel | Placebo Gel
Number analyzed (Participants) | 36 | 36
mm | 1.2 (2.9) | 19.2 (11.9)

3. Secondary Outcome: Neck Disability Index
Description: Neck Disability Index total score. Minimum = 0 "Best". Maximum = 50 "Worst"
Time Frame: 96h
Measure: Mean (Standard Deviation); unit: Total Score
Arm/Group | Diclofenac Diethylamine 1.16% Gel | Placebo Gel
Number analyzed (Participants) | 36 | 36
Total Score | 2.8 (3.0) | 14.6 (6.8)

ADVERSE EVENTS:
Arm/Group | Diclofenac Diethylamine 1.16% Gel | Placebo Gel
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 1/36
OTHER ADVERSE EVENTS (reported when occurring in more than 2.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diclofenac Diethylamine 1.16% Gel (N=36) | Placebo Gel (N=36)
Headache (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Preliminary agreement between Novartis Consumer Health and the investigator